CLINICAL TRIAL: NCT06400459
Title: Phase 1/2a, Proof-of-Concept, Multicenter, Parallel, Vehicle-Controlled, Double-Masked, Randomized Study Evaluating the Safety, Tolerability, and Efficacy of IVW-1001 Ophthalmic Eyelid Wipe in Subjects With Dry Eye Disease
Brief Title: IVW-1001 Phase 1/2 in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IVIEW Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVW-1001-CS-101
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Double-masked
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IVW-1001 0.1% (Experimental): IVW-1001 Ophthalmic Eyelid Wipe 0.1%
  Interventions: Drug: IVW-1001 Ophthalmic Eyelid Wipe 0.1%
- IVW-1001 0.2% (Experimental): IVW-1001 Ophthalmic Eyelid Wipe 0.1%
  Interventions: Drug: IVW-1001 Ophthalmic Eyelid Wipe 0.2%
- IVW-1001 Placebo (Placebo Comparator): Vehicle
  Interventions: Drug: IVW-1001 Placebo

INTERVENTIONS:
Drug: IVW-1001 Ophthalmic Eyelid Wipe 0.1% — IVW-1001 Ophthalmic Eyelid Wipe 0.1%
  Arms: IVW-1001 0.1%
Drug: IVW-1001 Ophthalmic Eyelid Wipe 0.2% — IVW-1001 Ophthalmic Eyelid Wipe 0.2%
  Arms: IVW-1001 0.2%
Drug: IVW-1001 Placebo — IVW-1001 Placebo
  Arms: IVW-1001 Placebo

SUMMARY:
Double-masked, dose-response, trial of IVW-1001 in subjects with dry eye disease.

DETAILED DESCRIPTION:
This is a randomized (1:1:1), multicenter, parallel, vehicle-controlled, double-masked study to evaluate the safety, tolerability, and efficacy of IVW-1001 Ophthalmic Eyelid Wipes in subjects with DED. Treatments will be IVW-1001 Ophthalmic Eyelid Wipe 0.2% (high dose), IVW 1001 0.1% (low dose), or IVW-1001 Ophthalmic Eyelid Wipe Placebo (vehicle). Subjects will participate in a 7-day, run-in period followed by a 28-daydosing period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of any gender at least 18 years of age at the Screening Visit
2. Able to voluntarily provide written informed consent to participate in the study
3. Able and willing to comply with all study procedures and restrictions, follow study instructions, and complete required study visits
4. Diagnosis of Dry Eye Disease (DED)

Exclusion Criteria:

1. Corneal fluorescein staining score of 4 using the NEI grading system
2. Intraocular pressure ≥23 mmHg
3. History of glaucoma or ocular hypertension in either eye requiring past or current medical or surgical intervention
4. Subjects with ocular inflammatory conditions (eg, conjunctivitis, keratitis, severe anterior blepharitis, etc.) not related to DED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Liang, PhD, Study Director — IVIEW Therapeutics Inc.
Locations (1):
- Houston Eye Associates, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVW-1001 0.1% | IVW-1001 0.2% | IVW-1001 Placebo
Started | 53 | 48 | 49
Completed | 53 | 48 | 49
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVW-1001 0.1% | IVW-1001 0.2% | IVW-1001 Placebo | Total
Number analyzed (Participants) | 53 | 48 | 49 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (11.19) | 63.5 (12.07) | 68.1 (11.43) | 65.1 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 39 | 113
  Male | 17 | 10 | 10 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 15 | 11 | 16 | 42
  White | 36 | 34 | 31 | 101
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 48 | 49 | 150
Unanesthetized Schirmer test (Study Eye) [Mean (Standard Deviation); unit: mm] — Unanesthetized measure of tear product using Schirmer strip (measured in mm of wetness)
  mm | 6.8 (1.98) | 6.1 (1.87) | 6.7 (1.92) | 6.5 (1.93)
Total Corneal Fluorescein Staining Score in the Study Eye (0, none to 20, severe) [Mean (Standard Deviation); unit: Score on a scale] — 0 (none) to 20 (severe)
  Score on a scale | 6.5 (1.37) | 6.8 (1.72) | 6.8 (1.48) | 6.7 (1.53)
Symptom Assessment in Dry Eye (SANDE): Frequency of Symptoms Score (0, none, to 100, severe) [Mean (Standard Deviation); unit: Score on a scale] — 0 (none) to 100 (severe)
  Score on a scale | 61.1 (23.3) | 62.6 (21.1) | 61.9 (23.0) | 61.8 (22.5)
Symptom Assessment in Dry Eye (SANDE): Severity of Symptoms Score [Mean (Standard Deviation); unit: Score on a scale] — 0 (none) to 100 (severe)
  Score on a scale | 54.9 (23.1) | 54.0 (20.2) | 55.0 (22.5) | 54.6 (21.9)
Symptom Assessment in Dry Eye (SANDE): Global Score [Mean (Standard Deviation); unit: Score on a scale] — 0 (none) to 100 (severe)
  Score on a scale | 57.5 (22.1) | 57.5 (23.1) | 57.5 (22.1) | 57.5 (22.4)

OUTCOME MEASURES:

1. Primary Outcome: Schirmer's
Description: Mean change from baseline in study eye in unanesthetized measure of tear product using Schirmer strip (measured in mm of wetness)
Time Frame: 29 Days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | IVW-1001 0.1% | IVW-1001 0.2% | IVW-1001 Placebo
Number analyzed (Participants) | 52 | 47 | 48
mm | 1.3 (6.40) | 2.1 (6.64) | 0.9 (5.24)

2. Secondary Outcome: Visual Acuity
Description: Mean change from baseline in best corrected visual acuity
Time Frame: 29 Days
Measure: Mean (Standard Deviation); unit: Logarithm of Minimum Angle of Resolution
Arm/Group | IVW-1001 0.1% | IVW-1001 0.2% | IVW-1001 Placebo
Number analyzed (Participants) | 53 | 48 | 49
Logarithm of Minimum Angle of Resolution | -0.007 (0.0739) | -0.013 (0.0625) | -0.014 (0.0728)

3. Secondary Outcome: Total Corneal Fluorescein Staining Score in the Study Eye
Description: Change from baseline in score on a scale (0 - none - to 20 - severe)
Time Frame: Week 4
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IVW-1001 0.1% | IVW-1001 0.2% | IVW-1001 Placebo
Number analyzed (Participants) | 53 | 48 | 49
Score on a scale | -1.65 (0.24) | -1.80 (0.25) | -1.10 (0.25)

4. Secondary Outcome: Symptom Assessment in Dry Eye (SANDE): Frequency of Symptoms Score
Description: Change from Baseline in the SANDE visual analog scale (0 - none to 100 - severe)
Time Frame: Week 4
Population: modified Intent to Treat
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IVW-1001 0.1% | IVW-1001 0.2% | IVW-1001 Placebo
Number analyzed (Participants) | 53 | 48 | 49
Score on a scale | -5.77 (2.91) | -23.57 (3.06) | -9.88 (3.08)

5. Secondary Outcome: Symptom Assessment in Dry Eye (SANDE): Severity of Symptoms Score
Description: Change from baseline in the SANDE visual analog scale (0 - none to 100 - severe)
Time Frame: 4 weeks
Population: modified intent-to-treat
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IVW-1001 0.1% | IVW-1001 0.2% | IVW-1001 Placebo
Number analyzed (Participants) | 53 | 48 | 49
Score on a scale | -8.73 (2.78) | -22.80 (2.93) | -12.55 (2.94)

6. Secondary Outcome: Symptom Assessment in Dry Eye (SANDE): Global Score
Description: Change from baseline in the SANDE visual analog scale (0 - none to 100 - severe)
Time Frame: 4 weeks
Population: Modified Intent to treat
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IVW-1001 0.1% | IVW-1001 0.2% | IVW-1001 Placebo
Number analyzed (Participants) | 53 | 48 | 49
Score on a scale | -7.11 (2.70) | -23.36 (2.84) | -11.16 (2.86)

ADVERSE EVENTS:
Time Frame: Week 4
Arm/Group | IVW-1001 0.1% | IVW-1001 0.2% | IVW-1001 Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/48 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 3/53 | 5/48 | 4/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVW-1001 0.1% (N=53) | IVW-1001 0.2% (N=48) | IVW-1001 Placebo (N=49)
Eye disorders (Eye disorders) | 3 (3) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators to collaborate with Sponsor on publication.

DOCUMENTS (2):
  • Study Protocol (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT06400459/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT06400459/SAP_001.pdf